CLINICAL TRIAL: NCT06347692
Title: Effect of Antigravity Treadmill Training on Pain, Gait Characteristics, and Function in Patients With Knee Osteoarthritis- A Randomized Controlled Trial
Brief Title: Effect of Antigravity Treadmill in Knee Osteoarthritis (AGTreadmill)
Acronym: AGTreadmill
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCBR-240/2024
Record Dates: First submitted 2024-02-27; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
Keywords: antigravity treadmill; osteoarthritis; gait characteristics; patient function
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: The study included 40 patients with knee osteoarthritis who were randomly assigned to one of two groups: the antigravity treadmill group (n=20) or the control group (n=20). For 12 weeks, the antigravity treadmill group received training on the Alter G treadmill (75% weight-bearing, 30 minutes per session, three times per week) combined with traditional physical therapy. During the same period, the control group received only traditional physical therapy. The Visual Analogue Scale, Walkway System, and the Western Ontario and McMaster Universities Arthritis Index were used to assess pain, spatiotemporal gait parameters, and patient function, respectively. All outcome measures were obtained pretreatment, post-treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were randomly assigned to either the antigravity treadmill group (n = 20) or the control group (n = 20 ) using an online randomization website (www.randomization.com). The control group received a conventional physical therapy program. The therapists responsible for measuring and assessing the outcomes remained blinded to the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): The control group received a conventional physical therapy program.
  Interventions: Other: physical therapy exercise program
- study group (Experimental): Conversely, in addition to the conventional physical therapy program provided to the control group, the antigravity treadmill group underwent antigravity treadmill training using the Alter G device.
  Interventions: Other: antigravity treadmill

INTERVENTIONS:
Other: antigravity treadmill — An Alter G treadmill (Alter G Pro 200, Alter G Inc, USA) was used to provide training to the patients in the antigravity treadmill group. The Alter G allows the patient to change their body weight from 20% to 100% in 1% increments. The air pressure inside the lower body positive pressure chamber can be adjusted from 0 to 2.0 kilopascal above atmospheric pressure. They are very comfortable to train in for long periods of time and have simple controls for adjusting body weight, speed, and inclination.
  Arms: study group
Other: physical therapy exercise program — Both groups received the same traditional physical therapy program for 12 weeks, three times a week, for 30 min each. The conventional physical therapy treatment consisted of acupuncture transcutaneous electrical nerve stimulation, Hot moist pack, Ultrasound and quadriceps setting
  Arms: control group

SUMMARY:
To date, the anti-gravity treadmill, as a representative method of lower body positive pressure treadmills, has been rarely reported for knee osteoarthritis rehabilitation.

Purpose: This study aims to evaluate the effect of antigravity treadmill training on pain, gait characteristics, and function in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
The study included 40 patients with knee osteoarthritis who were randomly assigned to one of two groups: the antigravity treadmill group (n=20) or the control group (n=20 ). For 12 weeks, the antigravity treadmill group received training on the Alter G treadmill (75% weight-bearing, 30 minutes per session, three times per week) combined with traditional physical therapy. During the same period, the control group received only traditional physical therapy. The Visual Analogue Scale, Walkway System, and the Western Ontario and McMaster Universities Arthritis Index were used to assess pain, spatiotemporal gait parameters, and patient function, respectively. All outcome measures were obtained pretreatment, post-treatment, and 3 months follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients should: (1) be ≥50 years old
* Patients have been diagnosed with mild to moderate osteoarthritis by a physician and confirmed by radiograph imaging (Kellgren & Lawrence grade 1-3)
* Patients complain of knee pain during the past 30 days when walking, squatting, and/or kneeling (the minimum level 3/10 on visual analogue scale before inclusion)
* Patients' body mass index greater than 30.

Exclusion criteria

* Patients were excluded if they have a history of ankle, knee, or hip injury or medical operation
* Have used knee injection for their knee osteoarthritis pain within the past year
* Have a history of other medical conditions that would interfere with walking
* Received physical therapy during the past 3 months for knee osteoarthritis
* Had any metabolic, pulmonary, neuromuscular, neurological, and/or autoimmune disease.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-07 (Estimated); Primary Completion 2024-04-20 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of patient pain | Pre and post 3 months intervention period
  The visual analogue scale is a reliable, valid, responsive, and frequently used pain outcome measure. It consists of a bidirectional 10 cm straight line with two labels, that is, "no pain" and "worst possible pain", located at either end of the line. Patients are instructed to draw a vertical mark on the line indicating their pain level.
Evaluation of gait parameters (step length) | Pre and post 3 months intervention period
  Gait parameters were measured using walkway System. The researcher assessed step length in centimeters
Evaluation of gait parameters (step time) | Pre and post 3 months intervention period
  Gait parameters were measured using walkway System. The researcher assessed step time in seconds
Evaluation of gait parameters (velocity) | Pre and post 3 months intervention period
  Gait parameters were measured using walkway System. The researcher assessed velocity which is measured in centimeter/second
Evaluation of patient function | Pre and post 3 months intervention period
  The Western Ontario and McMaster Universities Arthritis Index was used for assessing activities of daily living, functional mobility, gait, general health, and quality of life in patients with knee osteoarthritis. It has a total of 24 items and three subscales, namely pain (5 items), stiffness (2 items), and function (17 items), scored on a five-point ordinal scale, 0 - none, 1 - mild, 2 - moderate, 3 - severe, and 4 - extremely severe. Higher scores indicate worse pain, stiffness, and functional limitations.

IPD SHARING:
Plan to Share IPD: No